CLINICAL TRIAL: NCT05393687
Title: The Effect of Ankle Muscle Strengthening on Underwater Dolphin Kick Performance in Young Swimmers
Brief Title: Eccentric Strength Training of Ankle Joint Muscles in Swimming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DolphiKick
Record Dates: First submitted 2022-01-30; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Resistance Training
Keywords: swimming; resistance training; youth sports; elastic band; ankle

STUDY DESIGN:
Intervention Model Description: In order to examine the effect of strengthening exercises on performance amongst competitive young swimmers, a randomized controlled trial was undertaken. Swimmers were divided into two groups: Exercise (n=13) and the control groups (n=13). Both groups were assessed for 5-metre underwater swim time and ankle muscle strength before and after 8 weeks of normal swimming training. The exercise group received eccentric ankle strengthening exercises with an elastic band, in addition to their regular swimming training. Participants completed 24 exercises over 8 weeks, with 3 non-consecutive training sessions per week. Dynamic (2 minutes) and static stretching (2 minutes) exercises were performed as before the training session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eccentric exercise group (Experimental): 8 weeks of progressive eccentric ankle muscle strengthening program with elastic bands. Regular swimming training program five times a week.
  Interventions: Other: Eccentric exercise
- Control group (No Intervention): Regular swimming training program five times a week.

INTERVENTIONS:
Other: Eccentric exercise — progressive eccentric exercise with elastic band
  Arms: eccentric exercise group

SUMMARY:
This study was conducted to investigate the effectiveness of ankle muscle strengthening program of 8 weeks on the underwater dolphin kick performance in young swimmers. This study was a randomized controlled trial. Swimmers was divided in two groups; eccentric ankle muscle-strengthening exercises and control group. The outcome measures were strength of plantar flexors, dorsal flexors, internal rotators, external rotators and 5-meter underwater dolphin kick time.

DETAILED DESCRIPTION:
There is limited information on the effectiveness of ankle joint muscles in respect to the knee, hip, back and upper extremity muscles creating the propulsive forces for the feet to transfer the moment force towards water. Therefore, it is aimed to observe the effects of eccentric ankle muscle-strengthening exercises given by means of elastic bands on the Underwater Dolphin Kick performance of young swimmers.

ELIGIBILITY:
Inclusion Criteria:

* Having swimming training at least three times per week for the last year and using the proper UDK technique, which was assessed by the swimming trainer of the participants.

Exclusion Criteria:

* having any lower extremity injury or low back pain.

Ages: 84 Months to 155 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2016-10-09 (Actual); Study Completion 2016-10-09 (Actual)

PRIMARY OUTCOMES:
Underwater swim performance. | change in 5-meter underwater dolphin kick time in 8 weeks]
  5-meter underwater dolphin kick time measurement by using a chronometer.
Muscle Strength | change in ankle muscle strength in 8 weeks]
  Ankle muscle strength measurement (dorsal flexors, plantar flexors, internal rotators, external rotators) by using manual dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap İnal, Study Director — Istinye University
Locations (2):
- Turkey (Türkiye) (2):
  - Habibe Serap İnal, Şişli, Istanbul
  - Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istinye University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willems TM, Cornelis JA, De Deurwaerder LE, Roelandt F, De Mits S. The effect of ankle muscle strength and flexibility on dolphin kick performance in competitive swimmers. Hum Mov Sci. 2014 Aug;36:167-76. doi: 10.1016/j.humov.2014.05.004. Epub 2014 Jun 28. PMID 24984154
- [Background] von Loebbecke A, Mittal R, Fish F, Mark R. A comparison of the kinematics of the dolphin kick in humans and cetaceans. Hum Mov Sci. 2009 Feb;28(1):99-112. doi: 10.1016/j.humov.2008.07.005. Epub 2008 Nov 4. PMID 18986721
- [Background] Connaboy C, Naemi R, Brown S, Psycharakis S, McCabe C, Coleman S, Sanders R. The key kinematic determinants of undulatory underwater swimming at maximal velocity. J Sports Sci. 2016;34(11):1036-43. doi: 10.1080/02640414.2015.1088162. Epub 2015 Sep 14. PMID 26367778